CLINICAL TRIAL: NCT01589939
Title: Reduced PTV Margins for the Treatment of Prostate Cancer With IMRT Using Real-Time, State-of-the-Art Motion Tracking With the Calypso 4D Localization System: A Feasibility Study
Brief Title: Reduced Planning Target Volume (PTV) Margins for the Treatment of Prostate Cancer Using the Calypso 4D Localization System
Acronym: PTV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other)
Responsible Party: Principal Investigator, Dusten Macdonald, MD, MD, MC, Madigan Army Medical Center
Other Study IDs: W81XWH-08-2-0174, A-15214.1a; 207111 (Other: Madigan Army IRB)
Record Dates: First submitted 2012-04-26; First posted 2012-05-02 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer
Keywords: Reduced Planning Target Volume; radiation therapy; Calypso
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This prospective study evaluates the clinical utility of a novel real-time localization system allowing for smaller volumes of normal tissue to be included in radiation field and determines dosimetric parameters and adverse effect profiles of radiation therapy using this technology. Subjects will have beacon transponders implanted into the prostate to more precisely localize the position of the organ during radiation therapy. Hypothesis: 1. Treatment with highly targeted radiation therapy can be delivered in a daily treatment time consistent with routine clinical practice. 2. Highly targeted radiation therapy with reduced PTV margin will result in a significant decrease in rectal and bladder volume treated.

DETAILED DESCRIPTION:
This study will seek to establish the clinical feasibility of a novel real-time localization and tracking system for use of reduced PTV margins during intensity modulated radiation therapy (IMRT), which will allow treatment of smaller volumes of normal tissue during radiation therapy. Such a reduction in the PTV margins and the exposure of healthy tissue during treatment may allow for several future improvements in prostate radiotherapy including:

* decreased acute and chronic adverse effects with similar local tumor control
* dose escalation to achieve higher cure rates with similar adverse effects to standard dose treatment
* hypofractionation to shorten the time of, and lower the expense of, treatment without increased adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Low Risk: T1a, T1b, T1c, T2a; Gleason Score less than 7, PSA less than or equal to 10
* Intermediate Risk: T2b, T2c; Gleason Score less than or equal to 7, PSA less than or equal to 15
* Ability to comply with study schedule
* Age 40 or older
* Zubrod PS 0 or 1
* Signed informed consent

Exclusion Criteria:

* Node positive or metastatic prostate cancer
* Prior treatment of prostate cancer with surgery, chemotherapy, cryotherapy or brachytherapy
* History of prior pelvic radiotherapy
* History of abdominoperineal resection
* History of HIV infection
* History of chronic prostatitis or chronic cystitis
* History of bleeding disorder or any active anticoagulation (excluding ASA)
* PT or INR outside normal range for institution
* Active implanted devices such as cardiac pacemakers and automatic defibrillators.
* Prosthetic implants in the pelvic region that contain metal or conductive materials (eg., an artificial hip).
* Patients with maximum anterior-posterior separation through the torso minus the height of the center of the prostate greater than 17 cm (technical reason for Calypso System, see appendix 8).
* Prior history of androgen deprivation therapy has been deleted and these patients are allowed on study.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with localized prostate cancer for whom definitive radiation therapy is planned to the prostate only or prostate and seminal vesicle only, without ajuvant or neoadjuvant hormornal therpy will be referred by the radiation oncololgists and urologists.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Radiation therapy with reduced treatment margins can be adopted as feasible for routine clinical use | Approximately 8.5 weeks (43 fractions per pt.)
  During each radiation treatment fraction, therapists will record set up time, treatment time, total time and number of treatment interventions (repositioning/pausing) as well as the duration of the intervention caused by organ/target motion beyond planning target volume (PTV) margin using real time localization and tracking.

SECONDARY OUTCOMES:
Analyze dosimetric characteristics of treatment planning | usually within the first 2 weeks after beacon placement (done at simulation CT)
  Standard methods vs. reduced planning target volume expansions will be analyzed:
  1. Dose Volume Histogram (DVH), bladder and rectum
  2. Volume receiving 77.4Gy by the prescription dose (V77.4Gy), V70Gy, and V50Gy of bladder and rectum
Assess incidence of acute bladder and rectal toxicity | approximately 25 months (assessed prior to beacons are placed and then throughout treatment and follow-up)
  toxicity is based on the RTOG/NCI CTC and EPIC quality of life survey.

CONTACTS AND LOCATIONS:
Overall Officials: Dusten Macdonald, MD, Principal Investigator — Department of the Army
Locations (1):
- Madigan Healthcare System, Tacoma, Washington, United States